CLINICAL TRIAL: NCT02459470
Title: Utility of Stroke Volume Variation and Pulse Pressure Variation for Predicting Fluid Responsiveness in Chronic Renal Failure Patients Undergoing Kidney Transplantation
Brief Title: Stroke Volume Variation and Pulse Pressure Variation as Predictors of Fluid Responsiveness During Kidney Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: 2013-03-080; 2013-03-180 (Other: Samsung Medical Center)
Record Dates: First submitted 2015-05-14; First posted 2015-06-02 (Estimated); Last update posted 2015-06-02 (Estimated); Status verified 2012-12

CONDITIONS: Kidney Transplantation
Keywords: Fluid Responsiveness; Pulse Pressure Variation; Stroke Volume Variation
MeSH Terms: interventions — Hydroxyethyl Starch Derivatives; HES 130-0.4

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- SVV and PPV (Experimental): SVV(stroke volume variation): recorded using the Flotrac/Vigileo system (Edwards Lifesciences)
  PPV(pulse pressure variation): recorded using philips Intelivue MP70 monitors (Philips Medical System)
  Intervention: Other: Fluid loading using HES 130/0.4; voluven; Fresenius Kabi; Stans, Switzerland
  Interventions: Procedure: Fluid loading

INTERVENTIONS:
Procedure: Fluid loading — fluid loading was performed by using 7ml/kg of 6% hydroxyethyl starch within 10 min to all patients
  Other Names: HES 130/0.4; voluven; Fresenius Kabi; Stans, Switzerland

SUMMARY:
The aim pf this prospective study is to investigate the ability of stroke volume variation (SVV) and pulse pressure variation (PPV) to predict fluid responsiveness in patients undergoing kidney transplantation.

DETAILED DESCRIPTION:
Optimal intraoperative fluid management guided by central venous pressure (CVP), a traditional intravascular volume status indicator has been established to improve transplanted graft function during renal transplantation. Recently, stroke volume variation (SVV) and pulse pressure variation (PPV), dynamic preload indices derived from the arterial waveform are increasingly advocated as predictors of fluid responsiveness in anesthetized patients and critically ill patients. However, their usefulness in renal failure patients undergoing renal transplantation has not been investigated. Thus, the aims of this study is to investigate accuracy of SVV and PPV for predicting fluid responsiveness in patients undergoing kidney transplantation.

ELIGIBILITY:
Inclusion Criteria:

- chronic renal failure patients undergoing renal transplantation

Exclusion Criteria:

* patients with cardiac arrhythmia
* patients with reduced left ventricular function (EF < 40%)
* patients with valvular heart disease
* patients intracardiac shunt
* patients with pulmonary hypertension
* patients with extensive peripheral vascular disease
* patients with preoperative use of vasopressors or inotropics

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2012-12; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
stroke volume variation from Flo stroke volume variation from FloTrac/Vigileo system | within 5 minutes after fluid expansion
  predictable of stroke volume variation from FloTrac/Vigileo system for fluid responsiveness
pulse pressure variation from philips Intelivue MP70 monitor | within 5 minutes after fluid expansion
  predictable of pulse pressure variation from philips Intelivue MP70 monitor for fluid responsiveness

CONTACTS AND LOCATIONS:
Overall Officials: Gaab Soo Kim, M.D, Ph.D., Principal Investigator — Department of Anesthesiology and Pain medicie, Samsung Medical Center
Locations (1):
- Samsung Seoul Hospital, Samsung Medical Center, Seoul, South Korea